CLINICAL TRIAL: NCT04402242
Title: Impact of Nociceptive-Level (NOL) Intraoperative Guided Remifentanil Analgesia Versus Standard Clinical Care (SCC) for Elective Major Abdominal Surgery
Brief Title: Impact of NOL Index Intraoperative Guided Remifentanil Analgesia
Acronym: Eu-MultiNOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019_0051
Record Dates: First submitted 2020-04-20; First posted 2020-05-26 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Abdominal Surgery
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, single blinded interventional study with 2 parallel groups: standard clinical care (SCC group, control group) and NOL-guided analgesia (NOL guided analgesia group, interventional group), stratified by site
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "SCS" Group (Sham Comparator): Receiving anesthesia according to routine standard care, with the use of the "hidden" NOL (used to compare the data at the end of anesthesia with those of the classic BIS - without monitoring of the anesthesia by the NOL (without adjustment of treatments ))
  Interventions: Device: Bispectral index
- NOL Group (Experimental): Receiving anesthesia monitored by the NOL
  Interventions: Device: Bispectral index + NOL index

INTERVENTIONS:
Device: Bispectral index — Anesthesia monitoring
  Arms: "SCS" Group
Device: Bispectral index + NOL index — Anesthesia monitoring
  Arms: NOL Group

SUMMARY:
The Physiological Monitoring Device (PMD-200™) system is comprised of a monitor and a designated finger probe containing 4 sensors. The sensors included are Photoplethysmography (PPG), Galvanic Skin Response (GSR), Accelerometer for movement (ACC) and Thermistor for peripheral temperature (TMP).

The PMD-200 is intended to be used for assessing the nociception level in anesthetized patients.

The purpose of the study is confirmation of a reduction in the dosage of remifentanil allowed by the monitoring of nociception by the NOL which could open the way to a double control of the administration of anesthetic agents: control of the administration of hypnotics by the bispectral index (BIS) and control of the administration of opiate by the NOL.

DETAILED DESCRIPTION:
The PMD-200 continuous pain monitor is intended to be used for assessing changes in pain levels. The system monitors the physiological responses to pain using a relative pain index from 0-100, called the Nociception Level (NOL®) index. In the NOL index, 0 represents no nociception or pain and 100 represents high nociception or pain level.

The PMD-200 system consists of a monitor and a specific finger probe containing 4 sensors. The sensors included are Photoplethysmography (PPG), Galvanic Skin Response (GSR), Accelerometer for movement (ACC) and Thermistor for peripheral temperature (TMP).

The PMD-200™ is intended to be used for assessing the nociception level in anesthetized patients. The device is European Conformity (CE) marked and commercially available.

Meier et al. recently published a randomized trial involving 80 patients for major abdominal surgery, one group receiving routine care and the other NOL-guided analgesia. In the latter group, the remifentanil concentration was reduced when NOL values were below 10 or increased when NOL values were above 25 for at least 1 minute. In both groups, propofol was titrated to have bispectral index values between 45 and 55. Remifentanil administration was reduced in the NOL-guided group: 0.119 ± 0.033 vs 0.086 ± 0.032 μg.kg.min (p < 0.001). In the NOL- guided group, 2 out of 40 (5%) patients had hypotension (mean blood pressure less than 55 mm Hg) compared to 11 out of 40 (28%) in the control group (p = 0.006) and 16 out of 40 (40%) patients received vasoactive drugs vs 25 out of 40 (63%) (p = 0.044).

Previous results cover a small number of patients treated in a single center. The purpose of this study is to confirm this result within a multicenter study involving a larger group of patients. Confirmation of a reduction in the dosage of remifentanil allowed by the monitoring of nociception by the NOL will open the way to a double control of the administration of anesthetic agents: control of the administration of hypnotics by the bispectral index (BIS) and control of the administration of opiate by the NOL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* American Society of Anesthesiologists score (ASA) I, II or III stable
* Laparotomy or laparoscopy for major, planned, digestive, urological or gynecological surgery under total intravenous anesthesia (expected total duration > 90 minutes)
* Having sign an informed consent form prior to any study specific procedure
* Being covered by a national health insurance

Non-Inclusion Criteria:

* Pregnancy/lactation
* Patient with antiarrhythmic agents
* Patient with Central nervous system disorder
* Patient with veinous approach difficulties
* Patient at risk of difficult mask ventilation or difficult intubation
* Concomitant use of any type of anesthesia other than general anesthesia (epidural anesthesia, spinal anesthesia, wall block, pericatricial infiltration). Wall blocks and pericatricial infiltrations are allowed if they are carried out at the end of the intervention
* Allergy or intolerance to any of the study drugs
* Patient not understanding French language
* Being deprived of liberty or under guardianship

Exclusion Criteria:

* Patient requiring the administration of succinylcholine
* Patient with hemodynamic abnormality just before induction of anesthesia (mean arterial pressure < 65 mm Hg or > 110 mm Hg, heart rate < 45/min or > 90/min
* Concomitant use of any type of anesthesia other than general anesthesia (epidural anesthesia, spinal anesthesia, wall block, pericatricial infiltration). Wall blocks and pericatricial infiltrations are allowed if they are carried out at the end of the intervention
* Concomitant use of IV lidocaine or continuous ketamine (IV, SE) during anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Remifentanil consumption during maintenance | surgery day (D0)
  Remifentanil consumption during anesthesia maintenance in μg/kg/min

SECONDARY OUTCOMES:
Remifentanil consumption during induction | surgery day (D0)
  Remifentanil consumption during anesthesia induction in μg/kg/min
Propofol consumption during induction | surgery day (D0)
  Propofol consumption during anesthesia induction in μg/kg/min
Propofol consumption during maintenance | surgery day (D0)
  Propofol consumption during anesthesia maintenance in μg/kg/min
Proportion of patients with intraoperative hemodynamic abnormality in the NOL index group compared to standard care group during induction | surgery day (D0)
  A hemodynamic abnormality is defined as:
  * administration of a vasoactive agent (ephedrine, phenylephrine, norepinephrine, adrenaline, atropine)
  * and/or average blood pressure < 55 mmHg or < 60 mmHg or < 65 mmHg for any length of time
  * an/or a systolic blood pressure > 140 mmHg for any length of time
  * and/or a heart rate < 45 or > 90 /min
Proportion of patients with intraoperative hemodynamic abnormality in the NOL index group compared to standard care group during maintenance | surgery day (D0)
  Mean Blood pressure events during anesthesia inductio A hemodynamic abnormality is defined as:
  * administration of a vasoactive agent (ephedrine, phenylephrine, norepinephrine, adrenaline, atropine)
  * and/or average blood pressure < 55 mmHg or < 60 mmHg or < 65 mmHg for any length of time
  * an/or a systolic blood pressure > 140 mmHg for any length of time
  * and/or a heart rate < 45 or > 90 /min
Proportion of patients with intraoperative anesthetic abnormality in the NOL index group compared to standard care group during induction | surgery day (D0)
  An anesthetic abnormality is defined as:
  * a bispectral (BIS) index < 40 or > 60 for at least one minute
  * and/or a Burst Suppression Ratio (BSR) index > 10% during one minute
  * and/or a NOL index > 25 or < 10 for at least 2 minutes
Proportion of patients with intraoperative anesthetic abnormality in the NOL index group compared to standard care group during maintenance | surgery day (D0)
  An anesthetic abnormality is defined as:
  * a bispectral (BIS) index < 40 or > 60 for at least one minute
  * and/or a Burst Suppression Ratio (BSR) index > 10% during one minute
  * and/or a NOL index > 25 or < 10 for at least 2 minutes
Wake up time | surgery day (D0)
  delay between the end of Propofol or Sugammadex/Neostigmine and extubation
Intensity of pain in PACU (post-anesthesia care unit) | surgery day (D0)
  Morphine consumption in PACU (post-anesthesia care unit)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan LE GUEN, MD, Principal Investigator — Foch HOSPITAL
Locations (3):
- France (3):
  - Hôpital d'Instruction des Armées - Sainte-Anne, Toulon, Provence-Alpes-Côte d'Azur Region
  - Hopital d'Instruction des Armées de Bégin, Saint-Mandé, Saint Mandé
  - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meijer FS, Martini CH, Broens S, Boon M, Niesters M, Aarts L, Olofsen E, van Velzen M, Dahan A. Nociception-guided versus Standard Care during Remifentanil-Propofol Anesthesia: A Randomized Controlled Trial. Anesthesiology. 2019 May;130(5):745-755. doi: 10.1097/ALN.0000000000002634. PMID 30829658